CLINICAL TRIAL: NCT06724302
Title: The Accuracy of Ultrasound Assessment of the Thickening Fraction of the Diaphragm, Parasternal Intercostal, and Abdominal Expiratory Muscles for Predicting Weaning Outcomes in Mechanically Ventilated Patients
Brief Title: Ultrasound Assessment of the Thickening Fraction of the Respiratory Muscles for Predicting Weaning Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amer Bahir Soliman, Principal investigator, Tanta University
Other Study IDs: 36265MD308/11/24
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Weaning From Mechanical Ventilation
Keywords: diaghragm; Parasternal intercostal; Abdominal expiratory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The accuracy of ultrasound assessment of the thickening fraction of the diaphragm, parasternal intercostal, and abdominal expiratory muscles for predicting weaning outcomes in mechanically ventilated patients. A prospective observational study

DETAILED DESCRIPTION:
Mechanical ventilation is a widely used and important life-saving therapeutic approach in the intensive care unit. Nevertheless, it can lead to number of complications, including ventilator-associated lung injury , respiratory muscle dysfunction, and ventilator-associated pneumonia, which can increase healthcare expenses and unfavorable impact on patient outcomes. Prompt cessation of mechanical ventilation is crucial in the management of critically ill patients, however, timing is critical when determining if a patient can be successfully extubated as premature discontinuation of mechanical ventilation can lead to increased cardiovascular and respiratory stress, carbon dioxide (CO2) retention and hypoxemia with up to 25% of patients requiring reinstitution of ventilator support .

Several parameters have been used to predict weaning outcomes such as minute ventilation, maximum inspiratory pressure, tracheal airway occlusion, dynamic compliance and rapid shallow breathing index (RSBI), but none has shown great prognostic accuracy.

Critically ill patients frequently develop respiratory muscle dysfunction that may contribute to difficult and prolonged weaning from mechanical ventilation. Monitoring of the respiratory muscles function is therefore very useful during the weaning process The diaphragm is the principal respiratory muscle and diaphragmatic dysfunction is a common occurrence in critically ill patients. Therefore, diaphragmatic ultrasonography has been recently proposed as a simple, non-invasive, and bedside method to evaluate diaphragmatic function before any weaning attempt . However, it was highlighted that diaphragm ultrasound is not sufficient for predicting weaning outcomes . When diaphragmatic dysfunction occurs, the extra diaphragmatic respiratory muscles, such as parasternal intercostal muscles (7) and , the expiratory muscles of the abdomen are recruited.(8) Thus, exploring the value of extra diaphragmatic respiratory muscles in predicting weaning outcomes is appropriate . preliminary studies have found that parasternal intercostal and abdominal expiratory muscles' thickness and thickening fraction can be measured by ultrasonography which could provide additional information in the assessment of the respiratory function.

The aim of this study is to evaluate the accuracy of ultrasound assessment of the thickening fraction of the diaphragm, parasternal intercostal, and abdominal expiratory muscles for predicting weaning outcomes in mechanically ventilated patients.

Primary outcome:

The primary outcome of the study will be to:

- determine the accuracy of the thickening fraction of the diaphragm, parasternal muscles and abdominal expiratory muscles in predicting weaning outcome.

Secondary outcome:

The secondary outcome will be to estimate:

1. Cut-off values of the thickening fraction of the diaphragm, parasternal intercostal, and abdominal expiratory muscles to predict weaning outcomes.
2. Maximal inspiratory pressure.

This prospective observational study will be performed from January 2025 to December 2025 in the post-surgical intensive care unit (ICU) of Tanta University Hospitals. following approval from our institutional ethical committee.

All data of patients will be confidential with secret codes and private file for each patient, also an informed consent will be obtained from every patient's guardian. Any unexpected risk encountered during the study will be clarified to the ethical committee and to the patients' guardians on time.

Research results will be only used for scientific purposes. Disposal of waste materials will be done according to the infection control policy.

Inclusion criteria:

Patients will be enrolled if they are ≥18 years old, on invasive mechanical ventilation (MV) for more than 48 h and are eligible for first spontaneous breathing trial (SBT) after fulfilling all the following criteria:

1. Resolution or improvement of the disease leading to MV.
2. Adequate oxygenation, indicated by arterial oxygen partial pressure to inspired oxygen fraction (PaO2/FiO2) ≥ 200 mmHg, both with positive end-expiratory pressure (PEEP) ≤ 5 cmH2O and rapid shallow breathing index< 105.
3. Adequate pulmonary function, indicated by a RR<30 breaths/min with VT ≥5 mL/kg ideal body weight (IBW) and no significant respiratory acidosis with normal serum electrolytes.
4. Stable hemodynamics status, without or with minimal vasopressors
5. Conscious and cooperative patient
6. Absence of excessive tracheobronchial secretion (<3 times suction in the past 8 hours).
7. Effective cough reflex.

Exclusion criteria:

1. Pregnancy.
2. Presence of tracheostomy, pleural effusion, pneumothorax, pneumomediastinum, or hemothorax.
3. Presence of rib fractures.
4. Pre-existing cervical spinal injury, history or final diagnosis of neuromuscular disorders, and diaphragmatic paralysis or disorders
5. Use of neuromuscular blocking agents within 48 hours.
6. A distorted abdominal wall anatomy, or damage to the abdominal wall.
7. Patients with localized fluid collections in the abdomen, hernias, abdominal wall hematomas, inguinal masses, femoral hernias, abdominal surgeries.
8. BMI≥ 40
9. Patients with previously failed SBT

Sample size calculation:

The sample size calculation was performed using G.power 3.1.9.2 (Universitat Kiel, Germany). The sample size was calculated according to the sensitivity of thickening fraction of the diaphragm to predict weaning success expected to be between (60%-90%) according to previous studies. Based on the following considerations: 0.05 α error and 80% power of the study, allocation ration 1:1. Six cases were added to overcome dropout. Therefore, 80 patients will be allocated.

Continuous monitoring of the vital signs including: heart rate, non-invasive arterial blood pressure, electrocardiogram (ECG), oxygen saturation (Spo2), respiratory rate and temperature will be done and laboratory investigations including ABG will be evaluated before SBT. ABG will be repeated 30 minutes after the beginning of the trial.

All eligible patients will undergo an hour of (SBT) . SBT is conducted using pressure support ventilation (PSV), with a support pressure (PS) of 8 cmH2o, (PEEP) of 5 cmH2O, and FiO2≤ 50%.(2) Ultrasonographic examination using (PHILIPS-CX50, extreme edition, Philips, Finland) will be performed 15 min from the beginning of SBT on the right hemidiaphragm, the right parasternal intercostal and abdominal expiratory muscles. The ultrasound examination will be performed by an investigator blinded to the clinical outcomes and the average value of three consecutive measurements will be used for analysis.

Criteria for unsuccessful spontaneous breathing trials (if any one or more of the following are met).: anxiety, restlessness, excessive sweating, apparent paradoxical breathing, signs of respiratory distress; PaO2 below 50-60 mmHg, SpO2 below 90%; Pa CO2 greater than or equal to 50 mmHg; pH levels below 7.32,; respiratory rate (RR) exceeding 35 breaths/minute; heart rate (HR) exceeding 140 beats/minute; systolic blood pressure exceeding 180 mmHg, systolic blood pressure below 90 mmHg, and/or new-onset arrhythmias.

Ultrasound Measurements:

● Diaphragm ultrasound: A high frequency transducer will be placed vertical to the chest wall, at the eighth or ninth intercostal space, between the anterior axillary and the mid-axillary lines, to observe the zone of apposition of the muscle 0.5 to 2 cm below the costophrenic sinus. The diaphragm structure has three layers: two parallel echoic lines (the diaphragmatic pleura and the peritoneal membrane) and a hypoechoic structure between them (the muscle). The model will be then switched to the M-mode to measure the diaphragm thickness during breathing. Three consecutive measurements will be taken, and the average value will be recorded. The diaphragm thickening fraction (DTF) will be calculated using the formula: (thickness at end-inspiration - thickness at end-expiration) / thickness at end-expiration * 100%.

● Parasternal intercostal muscle ultrasound: A high frequency probe will be positioned between the 2nd and 3rd ribs on the right side of the sternum. The probe will be moved until the parasternal intercostal muscle become visible; then, it will be switched to the M-mode to measure the thickness of the parasternal intercostal muscle during respiratory cycles. Three consecutive measurements will be performed, and the average value will be recorded. The parasternal intercostal muscle thickness fraction (PIMTF) will be calculated by dividing the difference between the thickness at end-inspiration and end- expiration by the thickness at end-expiration, then multiplying by 100%.

● Abdominal expiratory muscle ultrasound: Ultrasound examination of rectus abdominis will be done by placing the linear probe horizontally about 2-3 cm above the umbilicus and 2-3 cm away from the midline. Ultrasound examination of the internal oblique, external oblique and transverses abdominis will be done by placing the linear probe horizontally at the anterior axillary line, approximately at the mid-point of the right costal margin and the iliac crest.(8) then, it will be switched to the M-mode to measure the thickness of the expiratory abdominal muscles. Thickening fraction of the expiratory abdominal muscles can be calculated as follows =(end-expiratory thickness-end-inspiratory thickness)/end-inspiratory thickness)×100%).(12) Patients will be divided into two groups according to the outcome of weaning. A successful weaning is defined as SB for >48 h following extubation. A failed weaning is defined as reinstitution of mechanical ventilation during or at the end of the SBT, reintubation within 48 h of extubation or the use of non-invasive ventilation within 48 h.

The following measurements will be recorded:

1. Demographic data as age, sex, body mass index, (APACHE II) score, concurrent diseases, reason for mechanical ventilation, and length of mechanical ventilation until SBT, will be recorded.
2. The thickening fraction of the diaphragm, parasternal intercostal muscle and abdominal expiratory muscles.
3. Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) for ultrasound derived measurements.
4. Maximal inspiratory pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be enrolled if they are ≥18 years old, on invasive mechanical ventilation (MV) for more than 48 h and are eligible for first spontaneous breathing trial (SBT) after fulfilling all the following criteria:

  1. Resolution or improvement of the disease leading to MV.
  2. Adequate oxygenation, indicated by arterial oxygen partial pressure to inspired oxygen fraction (PaO2/FiO2) ≥ 200 mmHg, both with positive end-expiratory pressure (PEEP) ≤ 5 cmH2O and rapid shallow breathing index< 105.
  3. Adequate pulmonary function, indicated by a RR<30 breaths/min with VT ≥5 mL/kg ideal body weight (IBW) and no significant respiratory acidosis with normal serum electrolytes.
  4. Stable hemodynamics status, without or with minimal vasopressors
  5. Conscious and cooperative patient
  6. Absence of excessive tracheobronchial secretion (<3 times suction in the past 8 hours).
  7. Effective cough reflex .Exclusion Criteria:

  <!-- -->

  1. Pregnancy.
  2. Presence of tracheostomy, pleural effusion, pneumothorax, pneumomediastinum, or hemothorax.
  3. Presence of rib fractures.
  4. Pre-existing cervical spinal injury, history or final diagnosis of neuromuscular disorders, and diaphragmatic paralysis or disorders
  5. Use of neuromuscular blocking agents within 48 hours.
  6. A distorted abdominal wall anatomy, or damage to the abdominal wall.
  7. Patients with localized fluid collections in the abdomen, hernias, abdominal wall hematomas, inguinal masses, femoral hernias, abdominal surgeries.
  8. BMI≥ 40
  9. Patients with previously failed SBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled if they are ≥18 years old, on invasive mechanical ventilation (MV) for more than 48 h and are eligible for first spontaneous breathing trial (SBT)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
determine the accuracy of the thickening fraction of the diaphragm, parasternal muscles and abdominal expiratory muscles in predicting weaning outcome. | 2 years
  Thickness of muscle during inspiration/thickness of muscle during expiration

SECONDARY OUTCOMES:
1. Cut-off values of the thickening fraction of the diaphragm, parasternal intercostal, and abdominal expiratory muscles to predict weaning outcomes. | 2 years
  mm.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiNino E, Gartman EJ, Sethi JM, McCool FD. Diaphragm ultrasound as a predictor of successful extubation from mechanical ventilation. Thorax. 2014 May;69(5):423-7. doi: 10.1136/thoraxjnl-2013-204111. Epub 2013 Dec 23. PMID 24365607